CLINICAL TRIAL: NCT01651741
Title: Effects of Seaweeds Combined With Probiotics on Intestinal Function of Healthy Subjects: a Randomized, Double-blind, Placebo-controlled, Waiting-list Clinical Trial
Brief Title: Effects of Seaweeds Combined With Probiotics on Intestinal Function of Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea Institute of Planning & Evalution for Technology of Food, Agriculture, Forestry & Fisherie (Other)
Responsible Party: Principal Investigator, Jae-Woo Park, Associate Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 911029-1
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: Intestinal Microbiota; Probiotics; Seaweed; Healthy Subject
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seaweed and Duolac7S (Experimental): Seaweed: Real Seaweed granule, Duolac7S: Real probiotics
  Interventions: Dietary Supplement: Seaweed and Duolac7S
- Seaweed and Duolac7S-P (Placebo Comparator): Seaweed: Real Seaweed granule, Duolac7S-P: Placebo probiotics
  Interventions: Dietary Supplement: Seaweed and Duolac7S-P

INTERVENTIONS:
Dietary Supplement: Seaweed and Duolac7S — Seaweed and probiotics is composed of seaweed and Duolac7S.
  Seaweed:
  1. Form: brown granule
  2. Dosage and frequency: 1 pack (3 g), 2 packs per day (30 min after morning, and evening meal)
  3. Duration: 4 weeks of treatment period
  Duolac7S:
  1. The probiotics, Duolac7S, consist of 7 bacteria.
  2. Ingredients: Lactobacillus acidophilus, L. plantarum, L. rhamnosus, Bifidobacterium breve, B. lactis, B. longum, Streptococcus thermophilus.
  3. Dosage and frequency: 1 capsule (5✕1,000,000,000 bacteria/capsule [7✕100,000,000 viable cells/strain]), 2 capsules per day (30 min after morning and evening meal)
  4. Duration: 4 weeks of treatment period
  Other Names: Seaweed and probiotics
  Arms: Seaweed and Duolac7S
Dietary Supplement: Seaweed and Duolac7S-P — Seaweed and probiotics is composed of seaweed and Duolac7S-P(Placebo Duolac7S).
  Seaweed:
  1. Form: brown granule
  2. Dosage and frequency: 1 pack (3 g), 2 packs per day (30 min after morning, and evening meal)
  3. Duration: 4 weeks of treatment period
  Duolac7S-P:
  Duolac7S placebo has the same form, color and flavor as experimental intervention (Duolac7S). The dosage, frequency and duration is also the same as experimental intervention (Duolac7S).
  Other Names: Seaweed and placebo probiotics
  Arms: Seaweed and Duolac7S-P

SUMMARY:
The aims of this study are to investigate the effect of seaweeds which is one of the main ingredients of Korean traditional food 'Kimchi' and probiotics on intestinal function of healthy subjects.

DETAILED DESCRIPTION:
Kimchi is one of the the typical and main foods in Korea. Seaweed is one of the important ingredient of Kimchi and has been known to have antiinflammatory, anticoagulant and antiadhesive effects. As seaweeds are fermented in order to make Kimchi, it can encourage beneficial probiotics to grow and lead to preventing digestive problems such as constipation and diarrhea.

In this trial, we are going to investigate the effect of combination of seaweeds and probiotics on intestinal function of healthy subject by evaluating intestinal microbiota. The trial is a randomized, double-blinded, placebo-controlled, 2-arm study. Forty patients with normal intestinal condition will be randomly assigned to one of the 2 groups consisting of Seaweed with real probiotics or Seaweed with placebo probiotics. The assigned treatments will last for 4 weeks and the follow-up period will be 2 weeks.

Four weeks of administration of seaweeds and probiotics is expected to increase the amount of beneficial microbiota and reduce that of harmful microbiota in intestine. we will also use questionnaires such as K-GSRS (Korean Gastrointestinal symptom rating scale), WHOQOL (The World Health Organization Quality of Life) - BREF and Assessment of bowel function scores (frequency, consistency, ease of passage - based on Bristol stool scale) to assess the change of digestive symptoms and the quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 - 75, with a elementary-school diploma or higher, must be literate
2. One who does not have any diseases or clinical symptoms related to digestive system
3. One whose every question of KGSRS is under 3 points
4. One who agree on not taking other therapies during the trial
5. During the past 5 yrs, no history of organic lesion proven by colonoscopy
6. One who agree on consent form

Exclusion Criteria:

1. Patients who have abdominal operation in the past (exception: appendectomy, caesarean section, tubal ligation, laparoscopic cholecystectomy, hysterectomy and abdominal wall hernia repair)
2. Patients who have history of serious diseases (cholangitis, pancreatitis, enteritis, ulcer, bleeding, cancer, etc.)
3. Before participating clinical trial, one who took over-the-count medication affecting GI motility
4. One who took antibiotics, herbal medicine or probiotics within 2 wks before participating the trial
5. Pregnant woman
6. One who disagree on the consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change of intestinal microflora (7 strains of Lactic acid bacteria) | Visit 1(0week), Visit 2(4week)
  1. To investigate the changes of intestinal microbes before and after experiment, feces should be collected.
  2. The feces will be analyzed by the method of DGGE (denaturing gradient gel electrophoresis - PCR of DNA).

SECONDARY OUTCOMES:
Daily assessment of bowel function scores | Visit 1(0week), Visit 2(4week), Visit 3(6week)
  1. The patients should write diaries of stool's frequency, consistency and ease of passage
  2. Frequency (number of defecation in a day)
  3. Consistency (judged by Bristol scale)
  4. Ease of passage
KGSRS (Korean gastrointestinal symptom rating scale) | Visit 1(0week), Visit 2(4week), Visit 3(6week)
  GSRS(Gastrointestinal symptom rating scale) is composed of 15 questions associated with various digestive problems such as abdominal pain, gastrointestinal reflux, indigestion, diarrhea and constipation.
  KGSRS, the Korean version of GSRS, reflects the language and sociocultural environment of Korea. The reliability and validity was confirm by Gwan et al.,2008.
WHOQOL (The World Health Organization Quality of Life) - BREF | Visit 1(0week), Visit 2(4week), Visit 3(6week)
  WHOQOL - BREF consists of 4 categories and 26 questions assessing various types of quality of life such as physical, psychological, social relationships and environment function.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Woo Park, KMD, PhD, Principal Investigator — Department of Internal Medicine, College of Oriental Medicine, Kyung Hee University, 1 Hoegi-dong, Dongdaemun-gu, Seoul 130-701, Republic of Korea
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, Gangdong-gu, South Korea

REFERENCES:
- [Derived] Jeong JH, Jo YN, Kim HJ, Jin DE, Kim DO, Heo HJ. Black soybean extract protects against TMT-induced cognitive defects in mice. J Med Food. 2014 Jan;17(1):83-91. doi: 10.1089/jmf.2013.3023. PMID 24456358
- [Derived] Ko SJ, Kim J, Han G, Kim SK, Kim HG, Yeo I, Ryu B, Park JW. Laminaria japonica combined with probiotics improves intestinal microbiota: a randomized clinical trial. J Med Food. 2014 Jan;17(1):76-82. doi: 10.1089/jmf.2013.3054. PMID 24456357
- See also: This is the URL of the site in which the clinical trial will be conducted. — http://www.khnmc.or.kr/